CLINICAL TRIAL: NCT02222558
Title: A Phase 2B Study to Determine the Dose Response Pharmacokinetics of TSX-002 (Testosterone) in Hypogonadal Males
Brief Title: Oral Testosterone for the Treatment of Hypogonadism in Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TesoRx Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT-006
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Hypogonadism
Keywords: hypogonadism; Gonadal Disorders; Endocrine System Diseases; Testosterone; Testosterone enanthate; Testosterone undecanoate; Testosterone 17 beta-cypionate; Methyltestosterone; Androgens; Hormones; Hormones,; Hormone Substitutes,; Hormone Antagonists; Physiological Effects of Drugs; Pharmacologic Actions; Therapeutic Uses; Anabolic Agents; dihydrotestosterone
MeSH Terms: conditions — Hypogonadism; Gonadal Disorders; Endocrine System Diseases | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Period 1: Single Dose (Experimental): Period 1: Each study subject will receive an escalating single dose of TSX-002 (60, 90, 120, 180, 240 mg), with a minimum 3 day wash-out between each of the 5 escalating doses. After completing the 240 mg dose, a 7 day wash-out period will occur prior to Period 2.
  Interventions: Drug: TSX-002
- Period 2: Two Times Daily Dosing 90 mg (Experimental): Period 2: Each study subject dose is 90 mg twice daily of TSX-002, fasted for 17 days.
  Interventions: Drug: TSX-002
- Period 3: Two Times Daily Dosing 120 mg (Experimental): Period 2: Each study subject dose is 90 mg twice daily of TSX-002, fasted for 17 days. On Day 15, a serum Testosterone level will be drawn and used to dose titrate and randomized to BID or TID (as eligible). The TSX-002 dose will be down or up titrated.
  Period 3: Begins Day 18 with the first adjusted TSX-002 dose administered fasted two times daily. The Testosterone level on Day 22 will be used to perform the final, TSX-002 dose adjustment.
  Interventions: Drug: TSX-002
- Period 3: Three Times Daily Dosing 90 mg (Experimental): Period 2: Each study subject dose is 90 mg twice daily of TSX-002, fasted for 17 days. On Day 15, a serum Testosterone level will be drawn and used to dose titrate and randomized to BID or TID (as eligible). The TSX-002 dose will be down or up titrated.
  Period 3: Begins Day 18 with the first adjusted TSX-002 dose administered fasted three times daily. The Testosterone level on Day 22 will be used to perform the final, TSX-002 dose adjustment.
  Interventions: Drug: TSX-002
- Period 3: Two Times Daily Dosing 180 mg (Experimental): Period 2: Each study subject dose is 90 mg twice daily of TSX-002, fasted for 17 days. On Day 15, a serum Testosterone level will be drawn and used to dose titrate and randomized to BID or TID (as eligible). The TSX-002 dose will be down or up titrated.
  Period 3: Begins Day 18 with the first adjusted TSX-002 dose administered fasted two times daily. The Testosterone level on Day 22 will be used to perform the final, TSX-002 dose adjustment.
  Interventions: Drug: TSX-002
- Period 3: Three Times Daily Dosing 120 mg (Experimental): Period 2: Each study subject dose is 90 mg twice daily of TSX-002, fasted for 17 days. On Day 15, a serum Testosterone level will be drawn and used to dose titrate and randomized to BID or TID (as eligible). The TSX-002 dose will be down or up titrated.
  Period 3: Begins Day 18 with the first adjusted TSX-002 dose administered fasted three times daily. The Testosterone level on Day 22 will be used to perform the final, TSX-002 dose adjustment.
  Interventions: Drug: TSX-002

INTERVENTIONS:
Drug: TSX-002 — TSX-002 are capsules with testosterone as the active ingredient.
  Other Names: Testosterone

SUMMARY:
Low testosterone is a condition that occurs when the body is unable to produce sufficient quantities of testosterone. The medical name for low testosterone is hypogonadism. Hypogonadism can be caused by many factors. Symptoms include: decrease in libido, lack of energy and mood swings. The goal of testosterone replacement therapy is to return testosterone levels to the normal range and relieve symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetic (PK) parameters of testosterone after administration of TSX-002 (easy to swallow testosterone capsules) to hypogonadal men. This will be determined by blood sampling at specified times during the study. The study is also intended to evaluate the PK parameters of the testosterone metabolite, dihydrotestosterone (DHT), as well as the safety and tolerability of TSX-002. The study consists of three (3) periods, for which TSX-002 will be taken orally at various doses. Study duration is approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic hypogonadal male subjects (Testosterone > 100 and <300 ng/dL, two separate 10 am samples one week apart),
* 18-70 years old,
* Willing and able to provide informed consent and to participate in all 3 periods of the study.
* BMI < 35 kg/m2.

Exclusion Criteria:

* Malabsorption conditions (e.g. history of cholecystectomy, Inflammatory Bowel Disease, Pancreatitis, Celiac disease, Sprue, Dumping syndrome, Bariatric surgery; Short bowel syndrome, Lactose intolerance);
* Alcoholics or substance abuse;
* Gastroparesis; IPSS (International Prostate Symptom score) > 19; PSA (prostate-specific antigen)> 4 ng/ml;
* Congestive Heart Failure, uncontrolled (NYHC >1);
* Uncontrolled sleep apnea;
* Topical or injectable testosterone replacement therapy (any kind including dehydroepiandrosterone (DHEA) and nutritional supplements) within past 4 weeks;
* Testopel excluded if within 2 years;
* Aveed excluded if within past 6 months;
* Hematocrit > 50.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, MD, Principal Investigator — San Diego Sexual Medicine
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned enrollment for this study was up to 28 subjects. The actual enrollment of the study was 25 subjects, all of whom were included in the safety and PK evaluable populations. This was a single-center study conducted at San Diego Sexual Medicine medical clinic. First patient screened 27Aug2014, FPE 05Sep2014, LPE 28Jan2015, LPLV 24Apr2015.
Pre-assignment Details: Period 1: Each study subject received 5 escalating single doses of TSX-002. Period 2: Each study subject dose was 90 mg BID of TSX-002, fasted for 17 days. On Day 15, a serum Testosterone level was drawn and used to determine eligibility for randomization to a further treatment group (BID vs. TID) or continuation in a BID treatment regimen.
Period: Period 1: Single Dose
Arm/Group | Period 1: Single Dose | Period 2: Two Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 120 mg | Period 3: Three Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 180 mg | Period 3: Three Times Daily Dosing 120 mg
Started | 25 | 0 | 0 | 0 | 0 | 0
Completed | 21 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0 | 0 | 0
Period: Period 2: Two Times Daily Dosing 90 mg
Arm/Group | Period 1: Single Dose | Period 2: Two Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 120 mg | Period 3: Three Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 180 mg | Period 3: Three Times Daily Dosing 120 mg
Started | 0 | 21 | 0 | 0 | 0 | 0
Completed | 0 | 21 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Period 1: Single Dose | Period 2: Two Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 120 mg | Period 3: Three Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 180 mg | Period 3: Three Times Daily Dosing 120 mg
Started | 0 | 0 | 4 | 1 | 8 | 8
Completed | 0 | 0 | 4 | 1 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects that began each defined period.
Groups:
- All Study Participants: Study participants start in Period 1 and proceed to Period 2 and then Period 3 Period 1: Each study subject will receive an escalating single dose of TSX-002 (60, 90, 120, 180, 240 mg), with a minimum 3 day wash-out between each of the 5 escalating doses. After completing the 240 mg dose, a 7 day wash-out period will occur prior to Period 2.
  Period 2: Each study subject dose is 90 mg twice daily of TSX-002, fasted for 17 days.
  Period 3: Begins Day 18 with the first adjusted TSX-002 dose administered fasted two times daily. The Testosterone level on Day 22 will be used to perform the final, TSX-002 dose adjustment.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 54.4 [31 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: Percentage of subjects with response to treatment within each period. Response to treatment was considered when Testosterone Cavg was within the physiological range of Testosterone concentration, i.e. 300 - 1050 ng/dL.
Time Frame: Cavg from samples at Period 1: post dose hrs 0,1,2,3,4,5,6,8,12,16,24; Period 2: hrs 0,2,3,4,5,6,8,12,14,15,16,17,18,20,24; Period 3 BID: hrs 0,2,3,4,5,6,8,12,14,15,16,17,18,20,24; Period 3 TID: hrs 0,2,3,4,5,6,8,10,11,12,13,14,16,18,19,20,21,22,24
Population: Subjects who received TSX-002 and provided PK concentrations for the protocol required 24 hour collection periods.
Measure: Number; unit: percentage of subjects
Arm/Group | Period 1: Single Dose | Period 2: Two Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 120 mg | Period 3: Three Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 180 mg | Period 3: Three Times Daily Dosing 120 mg
Number analyzed (Participants) | 25 | 21 | 4 | 1 | 8 | 7
percentage of subjects | 67 | 57 | 50 | 100 | 25 | 57.1

ADVERSE EVENTS:
Time Frame: 17 September 2014 (first subject Day 0) to 23 April 2015 (last subject visit). Adverse events presented were collected from start of drug treatment to discontinuation or completion of study participation.
Description: An AE could have been any unfavorable and unintended sign, symptom. Subjects were asked a question "How have you been feeling since you were last asked?" at all visits from Day 0 to Exit.
  Each sign or symptom was graded on a 3-point scale (mild, moderate, or severe).
Arm/Group | Period 1: Single Dose | Period 2: Two Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 120 mg | Period 3: Three Times Daily Dosing 90 mg | Period 3: Two Times Daily Dosing 180 mg | Period 3: Three Times Daily Dosing 120 mg
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/21 | 0/4 | 0/1 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/25 | 7/21 | 1/4 | 1/1 | 2/8 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Single Dose (N=25) | Period 2: Two Times Daily Dosing 90 mg (N=21) | Period 3: Two Times Daily Dosing 120 mg (N=4) | Period 3: Three Times Daily Dosing 90 mg (N=1) | Period 3: Two Times Daily Dosing 180 mg (N=8) | Period 3: Three Times Daily Dosing 120 mg (N=8)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug, due to muscle injury due to prolonged muscle compression. Lab abnormalities included acute renal failure secondary to rhabdomyolysis, hyperkalemia, high creatinine kinase, and high level of potassium.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Single Dose (N=25) | Period 2: Two Times Daily Dosing 90 mg (N=21) | Period 3: Two Times Daily Dosing 120 mg (N=4) | Period 3: Three Times Daily Dosing 90 mg (N=1) | Period 3: Two Times Daily Dosing 180 mg (N=8) | Period 3: Three Times Daily Dosing 120 mg (N=8)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (7) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At 60 days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy and allow Sponsor 60 days to review and comment and provide written permission prior to publication.